CLINICAL TRIAL: NCT00015210
Title: Efficacy of Nefazodone in Cocaine Dependent Subjects
Brief Title: Nefazodone in the Treatment of Cocaine Dependence and Depression - 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Dominic Ciraulo, Principal Investigator, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-5-0013-4; Y01-5-0013-4
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: Cocaine Use Disorders Dependence Depression
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — nefazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Nefazodone (Active Comparator): Nefazodone 100 mg tablet, titrated to a maximum of 200 mg administered twice daily by treatment day 10. Drug tapered over 7 days at the conclusion of the treatment period. Treatment was administered for 8 weeks.
  Interventions: Drug: Nefazodone; Behavioral: Psychosocial Treatment
- Matched Placebo Tablet (Placebo Comparator): Matched placebo tablet, titrated up to 2 tablets twice daily by day 10 and tapered over 7 days at the conclusion of the study. Treatment period lasted 8 weeks.
  Interventions: Drug: Nefazodone; Behavioral: Psychosocial Treatment

INTERVENTIONS:
Drug: Nefazodone
  Other Names: Serzone
Behavioral: Psychosocial Treatment — All subjects attended a weekly 1-hour therapy session during the 8 week treatment period.
  Other Names: Indivdual Manual-quided relapse prevention therapy; or Individual Dug Counseling

SUMMARY:
The purpose of this study is the use of Nefazodone in the treatment of cocaine dependence and depression comorbidity.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety and efficacy of nefazodone (Serzone ) in depressed cocaine dependent subjects. This is a hypothesis-testing study which will explore whether cocaine usage will be reduced in the nefazodone treatment group compared to a placebo control group.

ELIGIBILITY:
Inclusion Criteria:

DSM-IV diagnosis of cocaine dependence, Depression score of 12 or above and history of depression. Males and non-pregnant, non-nursing females 21-55 years of age.

Exclusion Criteria:

Axis I diagnosis other than substance use disorder, major depression, anxiety of dysthymic disorder. Physiological dependence on alcohol. Significant medical or neurological history. Abnormal UA, CBC or Chem 23 (LFT's may be up to 3 times normal). Enrollment in an opiate-substitution treatment program within 45 days of enrollment in the present study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 1997-02; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Urine benzoylecgonine (BE) concentration | Study Weeks Basekine to Week 8
  Natural log BE in urine samples collected weekly were analyzed for the baseline week and the subsequent 8 treatment weeks.

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | Baseline through Study Week 8
  HAM-D collected on a weekly basis.
Cocaine-Craving Scale | Baseline through Week 8
  CCS scores were collected on a weekly basis.
Adverse Events Self Report | Study Weeks 1 through 8
  Data for adverse events were collected on a weekly basis
Alcohol Drug Use Inventory | Baseline through Study Week 8
  Subjects were asked about the amount of cocaine consumed and the number of days in cocaine was used in the previous week, on a weekly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Dom Ciraulo, M.D., Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ciraulo DA, Knapp C, Rotrosen J, Sarid-Segal O, Ciraulo AM, LoCastro J, Greenblatt DJ, Leiderman D. Nefazodone treatment of cocaine dependence with comorbid depressive symptoms. Addiction. 2005 Mar;100 Suppl 1:23-31. doi: 10.1111/j.1360-0443.2005.00984.x. PMID 15730347